CLINICAL TRIAL: NCT04971642
Title: Ultrasound Imaging of Tooth-periodontium Complex Using an Innovative Intraoral Transducer
Brief Title: Intraoral Ultrasound Imaging of Tooth-periodontium Complex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Mitacs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00099721
Record Dates: First submitted 2021-04-30; First posted 2021-07-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Alveolar Bone Loss; Periodontitis
Keywords: ultrasound; periodontium
MeSH Terms: conditions — Alveolar Bone Loss; Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound scanning (Experimental): The subjects recruited are existing patients of the Orthodontic Clinic - Oral Health Clinic-Dentistry, University of Alberta. An intraoral ultrasound scanning will be done on the buccal side of the upper and lower incisor/canine/premolar/molar teeth for a total of sixteen (16) teeth (four(4) teeth in each of the four quadrants) of these subjects.
  The ultrasound scans will be done separately by a research assistant not involved in patient care. The whole procedure for ultrasound scanning and data storage will take about 25-30 min including 3-5 min preparation time and 22-25 min of data acquisition and storage time.
  Interventions: Device: Intraoral ultrasound

INTERVENTIONS:
Device: Intraoral ultrasound — Intraoral ultrasound scanning of the periodontium complex

SUMMARY:
Misaligned teeth are very common in the population and are commonly known as malocclusion. This happens when the upper teeth do not align properly with the lower teeth. It can lead to difficulty in jaw movement, chewing, speech, and gum disease. Correction of malocclusion requires orthodontic (braces) treatment. Currently, the imaging technique known as cone-beam computed tomography (CBCT) has been routinely used in orthodontic diagnosis and treatment planning for patients with malocclusion. Although CBCT provides better information than conventional dental X-rays, it typically delivers more harmful radiation to the patients. This is especially important as radiation from repeated X-ray imaging during dental monitoring visits can be cumulative.

Ultrasound is commonly used in medical imaging. The ultrasound method is non-invasive, cost-effective, and free of ionizing radiation. The application of ultrasound has been investigated in many fields in Dentistry. We plan to evaluate the ability of intra-oral ultrasound to see the bone and gingiva around the tooth for patients under orthodontic treatment. If ultrasound is found to be a reliable tool in imaging the tooth-gum complex, children and adolescents will benefit immensely from the decreased radiation risks and reduced cancer rate.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to investigate a intraoral ultrasound to image the tooth-periodontium complex that is an alternative to ionizing radiation CBCT imaging.

Hypothesis:

Ultrasound imaging is a radiation-free alternative to image tooth-periodontium complex.

Justification:

Straight teeth and a healthy smile is paramount to an individual's well-being. Malocclusion (crowding of teeth) is the third most common dental anomaly according to the World Health Organization(WHO). The severity of malocclusion can cause difficulty in jaw movement, chewing, speech, and high susceptibility to gum disease. Correction of malocclusion problems requires comprehensive orthodontic treatment. CBCT imaging for orthodontic diagnosis and treatment planning has increased of late due to its inherent advantages over the traditional 2D planar cephalometric and panoramic radiography. These include the advantage of having 3D capabilities to view images with no superimposition or magnification errors. This is especially significant in detecting bony dehiscence and fenestration associated with orthodontic treatment. The presence of these defects decreases bony support to the teeth, which compounded with plaque-induced inflammation, can be detrimental to the health of the teeth during orthodontic tooth movement. CBCT image typically delivers much higher radiation than conventional dental radiographs. Orthodontic patients, mostly children, are increasingly susceptible to deleterious effects of ionizing radiation due to the accumulated radiation dose from repeated monitoring visits. Hence new imaging modalities such as ultrasound have been researched as a radiation-free alternative to CBCT imaging. The ultrasound technique uses echoes of mechanical waves and the acoustic properties of the target to produce an image non-invasively. The characteristics of the returning echoes are mainly governed by the elastic 'properties of the transmitting medium and the acoustic impedance contrast of the interface between the target and the surrounding medium. For decades, medical ultrasound has mainly been used to image soft tissues. Although the use of ultrasound in dentistry focused more on imaging dental hard tissues, most recently, its use has been expanded to image periodontal soft and hard structures. Although the interest in using ultrasound in dentistry is increasing, research on the use of ultrasound to study tooth-periodontal tissues is limited.

Objectives:

The objective of this study is to determine the validity and reliability of an intra-oral ultrasound technique in a clinical setting by comparing the ultrasound measurements with those of the clinical standard CBCT imaging.

Research Method/Procedures:

Participant recruitment:

60 orthodontic participants in the age group of 10-60 years old will be recruited for the study for over a year. This population group is screened and recruited from the patients seen at the Orthodontic Clinic in the Oral Health Clinic - Department of Dentistry based on the inclusion and exclusion criteria. Each subject will have diagnostic records taken as part of routine orthodontic diagnosis and treatment planning. These records include extraoral and intraoral photos, digital models, and CBCT imaging. In addition to routine diagnostic records, ultrasound scanning of the mandibular and maxillary incisor, canine, premolar, and molar teeth for a total of sixteen (16) teeth (four (4)teeth in each of the four quadrants) will be performed after obtaining informed consent from patients and their guardians. Following diagnostic records, all subjects will undergo orthodontic treatment for correction of their malocclusion by either a licensed orthodontic faculty member or an orthodontic resident under the supervision of a licensed orthodontist at Kaye Edmonton Dental Clinic, University of Alberta.

Procedures:

Ultrasound Scanning:

The ultrasound scanner used is a handheld medical diagnostic system that has a Clarius platform (ClariusMobile Health, Richmond, Canada, Device ID: 1012444 and DeviceIdentifier 99-02-00046

) and a DenSonics DSI-1 intraoral 20 MHz array transducer (DenSonics Imaging Inc, Edmonton, Canada) to be used off-label (Health Canada has not approved yet).

All ultrasound scans will be done by the same research assistant after training. This research assistant has no involvement in the patient's care. The ultrasound imaging will be performed on the maxillary and mandibular(again 16 teeth per patient will be imaged - incisor/canine/premolar/molar in each of the four dental quadrants). The tooth-periodontium complex will be imaged.

The probe will be isolated for infection control using a plastic wrap and will be positioned intraorally with a gel pad separating the ultrasound transducer and the targeted tooth-periodontium structures, with the long axis of the probe in alignment with the longitudinal axis of the tooth. On average, it takes about 1-2 minutes to perform a single scan, and we estimate a total of 25 minutes to perform scans on all the teeth in a single individual. The saved data will be exported to a desktop computer for data analysis and measurements using in-house developed MATLAB codes.

Plan for Data Analysis:

Outcome measures:

The following five distance, thickness, or localization parameters will be measured linearly on ultrasound images for further analysis and comparison: (1) gingival margin- cementoenamel junction, (2) cementoenamel junction - alveolar bone crest, (3) gingival thickness at the alveolar bone crest, (4) alveolar bone thickness at the crest and (5) localization of cementoenamel junction. Measurements of the above five parameters will be performed by four raters in the ultrasound images. All the raters will be blinded for data processing and measurement. To test intra-rater reliability, each rater will conduct the measurement three times with one week apart between measurements to avoid bias. Three of the measurements: (2) cementoenamel junction - alveolar bone crest, (4) alveolar bone thickness at the crest and (5) localization of cementoenamel junction will be identified in both CBCT and ultrasound images and compared.

Statistical analysis:

Descriptive statistics will be presented as Mean±SD. Quality control of the data will be done by scatter plots to detect outliers. We will consider three assessments: Intra-rater reliability, inter-rater reliability, and agreement between the two methods. The intra- and inter-rater reliabilities will be assessed by intra-class correlation coefficients (ICC(2,1)) using a 2-way random model and absolute agreement with a 95% confidence interval. Correlation and the Bland-Altman plot will be used to assess the agreement between CBCT and ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be recruited to the Orthodontic Clinic-Oral Health Clinic at the Department of Dentistry - University of Alberta based on the following inclusion criteria:

  1. Males or females in the age group of 10-60 years old
  2. Individuals with permanent dentition
  3. Dental malocclusion with mild to moderate crowding
  4. Individuals undergoing CBCT imaging as part of Orthodontic diagnostic records Individuals in the age group of 10-60 years would have a full complement of permanent teeth erupted which will help standardize the research methodology to prevent an error in data acquisition, caused by the overlap of dental tissue in the mixed dentition period.

Exclusion Criteria:

* Participants with missing permanent teeth, gingival recession (below CEJ), severe crowding, or a history of corrective orthodontics will be excluded. Any co-factors (previous orthodontic treatment) that might influence the ultrasound findings, will be excluded. Participants with unfavorable oral hygiene will be excluded due to the ambiguity associated with data acquisition in an inflamed periodontium. Also, participants presenting with craniofacial syndromes will be excluded due to the factors related to changes in craniofacial anatomy (maxilla-mandible anatomy)

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Distance from alveolar bone crest to the cemento-enamel junction | through study completion, an average of 1 year
  It is the linear measurement distance in millimeters (mm) from the alveolar bone crest to the cemento-enamel junction anatomical structures observed in the Ultrasound image. It will be evaluated using an image software.
Distance from cemento-enamel junction to the gingival margin | through study completion, an average of 1 year
  It is the linear measurement distance in millimeters (mm) from the cemento-enamel junction to the gingival margin observed in the Ultrasound image. It will be evaluated through an image software.
Gingival thickness | through study completion, an average of 1 year
  It is the linear measurement of the thickness of gingival tissue at the alveolar bone crest level in millimeters (mm) observed in the Ultrasound image. It will be evaluated using an image software
Alveolar bone thickness | through study completion, an average of 1 year
  It is the linear measurement of the alveolar bone thickness at the alveolar bone crest level in millimeters (mm) observed in the Ultrasound image. It will be evaluated using an image software.
Cemento-enamel junction identification | through study completion, an average of 1 year
  The Identification of the cemento-enamel junction will be done by adding a point to this anatomical structure in the ultrasound image. It will be evaluated using an image software

CONTACTS AND LOCATIONS:
Overall Officials: Fabiana Marques, PhD, Principal Investigator — University of Alberta
Locations (1):
- Oral Health Clinic, 8th Floor, Kaye Edmonton Dental Clinic., Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Data won't be shared for confidentiality reasons

REFERENCES:
- [Background] Nguyen KCT, Duong DQ, Almeida FT, Major PW, Kaipatur NR, Pham TT, Lou EHM, Noga M, Punithakumar K, Le LH. Alveolar Bone Segmentation in Intraoral Ultrasonographs with Machine Learning. J Dent Res. 2020 Aug;99(9):1054-1061. doi: 10.1177/0022034520920593. Epub 2020 May 11. PMID 32392449
- [Background] Nguyen KT, Le LH, Kaipatur NR, Zheng R, Lou EH, Major PW. High-Resolution Ultrasonic Imaging of Dento-Periodontal Tissues Using a Multi-Element Phased Array System. Ann Biomed Eng. 2016 Oct;44(10):2874-2886. doi: 10.1007/s10439-016-1634-2. Epub 2016 May 9. PMID 27160674
- [Background] Nguyen KC, Le LH, Kaipatur NR, Major PW. Imaging the Cemento-Enamel Junction Using a 20-MHz Ultrasonic Transducer. Ultrasound Med Biol. 2016 Jan;42(1):333-8. doi: 10.1016/j.ultrasmedbio.2015.09.012. Epub 2015 Nov 3. PMID 26546266
- [Background] Nguyen KT, Pacheco-Pereira C, Kaipatur NR, Cheung J, Major PW, Le LH. Comparison of ultrasound imaging and cone-beam computed tomography for examination of the alveolar bone level: A systematic review. PLoS One. 2018 Oct 3;13(10):e0200596. doi: 10.1371/journal.pone.0200596. eCollection 2018. PMID 30281591